CLINICAL TRIAL: NCT04920370
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study of Subcutaneous and Intravenous ALXN1720 With and Without rHuPH20 in Healthy Subjects
Brief Title: Study of Subcutaneous and Intravenous ALXN1720 With and Without rHuPH20 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN1720-HV-101; 2018-004500-19 (EudraCT Number)
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: ALXN1720; Safety; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ALXN1720 Single Dose SC (Experimental): Participants will receive a single dose of ALXN1720 SC.
  Interventions: Drug: ALXN1720 SC
- ALXN1720 Multiple Dose SC (Experimental): Participants will receive multiple doses of ALXN1720 SC.
  Interventions: Drug: ALXN1720 SC
- ALXN1720 Single Dose SC + rHuPH20 (Experimental): Participants will receive a single dose of ALXN1720 SC in combination with rHuPH20.
  Interventions: Drug: ALXN1720 SC; Drug: rHuPH20
- ALXN1720 Single Dose IV (Experimental): Participants will receive a single dose of ALXN1720 IV.
  Interventions: Drug: ALXN1720 IV
- Placebo (Placebo Comparator): Participants will receive Placebo SC or Placebo IV according to their assigned cohort.
  Interventions: Drug: Placebo SC; Drug: Placebo IV

INTERVENTIONS:
Drug: ALXN1720 SC — ALXN1720 will be administered via SC route.
  Arms: ALXN1720 Multiple Dose SC; ALXN1720 Single Dose SC; ALXN1720 Single Dose SC + rHuPH20
Drug: ALXN1720 IV — ALXN1720 will be administered via IV route.
  Arms: ALXN1720 Single Dose IV
Drug: rHuPH20 — rHuPH20 will be administered via SC route.
  Arms: ALXN1720 Single Dose SC + rHuPH20
Drug: Placebo SC — Placebo will be administered via SC route.
  Arms: Placebo
Drug: Placebo IV — Placebo will be administered via IV route.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of ALXN1720 administered subcutaneously (SC) or intravenously (IV).

DETAILED DESCRIPTION:
Participants will be randomized in a 3:1 ratio to receive the active treatment or placebo.

The study will be conducted in healthy adult participants, including participants of Japanese descent.

ELIGIBILITY:
Inclusion Criteria:

* Body weight within 50 to 90 kilograms (kg), inclusive, and body mass index within the range of 18 to 29.9 kg/meter squared, inclusive.
* Willing to follow protocol-specified contraception guidance while on treatment and for 6 months after the last dose of study treatment.
* Vaccination with tetravalent meningococcal conjugate vaccine and serogroup B meningococcal vaccine.
* No clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory evaluation.
* For the cohorts with Japanese participants, parents and grandparents must both be Japanese, and participants must have resided for less than 5 years outside of Japan.

Exclusion Criteria:

* Current or recurrent disease that could affect clinical assessments or clinical laboratory evaluations.
* History of complement deficiency or complement activity below the reference range.
* Female participants who are breastfeeding.
* Immunization with a live-attenuated vaccine 28 days prior to dosing on Day 1 or planned vaccination during the course of the study. Immunization with inactivated or recombinant influenza vaccine, or nucleoside-modified messenger ribonucleic acid or recombinant COVID-19 vaccine is permitted.
* Current tobacco smoking, history of illicit drug abuse, or history of significant alcohol abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent and Serious Adverse Events (TEAEs, SAEs) | Up to 176 days following the first day of dosing

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of ALXN1720 SC, ALXN1720 SC/rHuPH20, and ALXN1720 IV | Up to 176 days following the first day of dosing
Area Under The Concentration-time Curve (AUC) of ALXN1720 SC, ALXN1720 SC/rHuPH20, and ALXN1720 IV | Up to 176 days following the first day of dosing
Change from Baseline in Serum Concentrations of Free Complement Component 5 (C5) | Baseline, 176 days following the first day of dosing
Change from Baseline in Serum Concentrations of Total C5 | Baseline, 176 days following the first day of dosing
Change from Baseline in Ex Vivo Chicken Red Blood Cell (cRBC) Hemolysis Activity | Baseline, 176 days following the first day of dosing
Incidence of Antidrug Antibodies (ADAs) to ALXN1720 | Up to 176 days following the first day of dosing
Absolute Bioavailability of ALXN1720 | Up to 176 days following the first day of dosing
  The absolute bioavailability for ALXN1720 SC will be defined by the ratio of the geometric means for AUC for ALXN1720 SC over ALXN1720 IV after a single dose.
Comparison of Incidence of TEAEs and SAEs Between Healthy Non-Japanese Participants and Participants of Japanese Descent | Up to 176 days following the first day of dosing
Comparison of Cmax of ALXN1720 SC, ALXN1720 SC/rHuPH20, and ALXN1720 IV Between Healthy Non-Japanese Participants and Participants of Japanese Descent | Up to 176 days following the first day of dosing
Comparison of AUC of ALXN1720 SC, ALXN1720 SC/rHuPH20, and ALXN1720 IV Between Healthy Non-Japanese Participants and Participants of Japanese Descent | Up to 176 days following the first day of dosing
Comparison of Change from Baseline in Serum Concentrations of Free C5 Between Healthy Non-Japanese Participants and Participants of Japanese Descent | Baseline, 176 days following the first day of dosing
Comparison of Change from Baseline in Serum Concentrations of Total C5 Between Healthy Non-Japanese Participants and Participants of Japanese Descent | Baseline, 176 days following the first day of dosing
Comparison of Change from Baseline in Serum Concentrations in Ex Vivo cRBC Hemolysis Activity Between Healthy Non-Japanese Participants and Participants of Japanese Descent | Baseline, 176 days following the first day of dosing
Comparison of ADAs to ALXN1720 Between Healthy Non-Japanese Participants and Participants of Japanese Descent | Up to 176 days following the first day of dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, London, United Kingdom